CLINICAL TRIAL: NCT00006253
Title: Family Home Care for Cancer - A Community-Based Model
Brief Title: Pain and Fatigue Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Barbara Given, Associate Dean of Research, University Distinguished Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01CA079280 (NIH)
Record Dates: First submitted 2000-09-11; First posted 2004-03-08 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Carcinoma
Keywords: symptom management; cancer; chemotherapy treatment; Behavioral Research; Physiological Effects of Drugs; Clinical Trial, Phase II
MeSH Terms: conditions — Carcinoma; Neoplasms | interventions — Nurses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse (Experimental): Receives symptom management assistance from an oncology nurse via the telephone
  Interventions: Behavioral: Nurse
- Non-nurse coach (Experimental): Receives symptom management assistance from a non-nurse coach via telephone
  Interventions: Behavioral: Non-nurse coach

INTERVENTIONS:
Behavioral: Nurse — Receives 6 telephone calls over 8 weeks from an oncology nurse to assist with symptom management
  Arms: Nurse
Behavioral: Non-nurse coach — Receives 6 telephone calls over 8 weeks from a non-nurse coach to assist with symptom management
  Arms: Non-nurse coach

SUMMARY:
Patients with advanced cancer who are undergoing chemotherapy and who report pain and fatigue at intake in the past 24 hours or at a level 2 or higher of pain or fatigue at a 3 or higher on a 10-point scale will be assigned randomly to an 8-week, 6-contact self management attention control (SMAC) intervention, or to a 8-week, 6-contact experimental patient intervention for management of symptoms and support (PIMSS) targeted toward symptom management, reducing impact on physical role and social functioning and emotional distress. Both groups will continue to receive conventional cancer care.

When compared with the self-management attention control intervention, patients exposed to the experimental intervention will report statistically significant positive effects on the following:

1. The primary outcome--total number of symptoms reported;
2. The secondary patient outcomes--reduced deterioration in physical role impact and social functioning, emotional distress, levels of communication with caregiver about care, and communication and satisfaction with provider care; and
3. Caregiver outcomes--greater involvement in symptom management, increased mastery of the caregiving process, reduced levels of depression and burden.

DETAILED DESCRIPTION:
GOAL: The primary goal of this research is to test a symptom management intervention, delivered by nurses with special training, using a stepped-care approach targeted toward pain and fatigue, followed by fifteen other prevalent cancer symptoms. Second goals are to improve physical and social functioning, lower emotional distress, and improve communication with family caregiver in symptom management, and assist them to reduce their levels of depression and burden. This research is funded through a grant from the National Cancer Institutes, and builds upon the Family Care Research Team's program of supportive cancer-care research.

OUTCOMES: This study tests a stepped-approach intervention to determine if it improves symptom outcomes, especially pain and fatigue. Secondary outcomes addressed by the intervention are physical role impact, social functioning, and emotional distress. These outcomes can have significant impact on patients and family caregivers' well-being as patients undergo chemotherapy. The shorter, more intense intervention corresponds to changes int he clinical management of cancer patient with more intense, shorter chemotherapy treatments; therefore, this intervention will be more easily translatable to the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* solid tumor cancer diagnosis
* receiving chemotherapy treatment
* advanced cancer
* family caregiver

Exclusion Criteria

* Emotional or psychology disorder for which patient is receiving treatment
* does not speak English
* does not have access to a telephone
* difficulty hearing on the telephone

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2003-03; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Primary patient outcome
  Lower reported severity of symptoms

SECONDARY OUTCOMES:
Secondary Patient Outcomes
  Reduced deterioration in physical role impact and social functioning, emotional distress, levels of communication with caregiver about care and communication, and satisfaction with provider care

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Given, PhD, RN, FAAN, Study Chair — Breslin Cancer Center at Ingham Regional Medical Center
Locations (1):
- Michigan State University, East Lansing, Michigan, United States